CLINICAL TRIAL: NCT03127111
Title: The Identification, Validation and Implementation of Molecular Markers to Predict Response to Fluorouracil-based Adjuvant Chemotherapy in Stage III Colorectal Cancer Patients - Prospective Clinical Observational Study
Brief Title: Genetic and Epigenetic Determinants of Response to Fluorouracil-based Adjuvant Chemotherapy in Patients With Stage III Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Tao Fu, Head of Department of GI Surgery II, Renmin Hospital of Wuhan University
Other Study IDs: GEDEREFAC-CRC
Record Dates: First submitted 2017-04-16; First posted 2017-04-25 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Stage III Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Gene Expression Profiling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, serum, tumor tissue, normal colorectal tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adjuvant chemotherapy: Samples from patients with stage III colorectal cancer who are going to receive fluorouracil-based adjuvant chemotherapy will be used for gene mutations analysis, gene methylation analysis, gene expression analysis, SNP analysis, and protein expression analysis.
  Interventions: Genetic: Gene mutations analysis; Genetic: Gene methylation analysis; Genetic: Gene expression analysis; Genetic: SNP analysis; Genetic: Protein expression analysis

INTERVENTIONS:
Genetic: Gene mutations analysis — Genomic DNA extracted from paired fresh-frozen tumor and normal tissues is used for KRAS mutations, BRAF mutations, PIK3A mutations, and EGFR mutations, etc., by sequencing and for MSI analysis by PCR and capillary electrophoresis.
Genetic: Gene methylation analysis — Genomic DNA extracted from paired fresh-frozen tumor and normal tissues is used for specific gene methylation or CIMP status analysis by MethyLight or bisulfite sequencing. Whole-genome bisulfite sequencing will be used to identify novel candidate set of predictive markers.
Genetic: Gene expression analysis — RNA extracted from paired fresh-frozen tumor and normal tissues or serum is used for specific gene expression analysis by real-time reverse-transcription PCR (RT-qPCR). RNA-seq will be used to identify novel candidate set of predictive markers.
Genetic: SNP analysis — Genomic DNA extracted from serum is used for specific SNP analysis by using sequencing. GWAS with SNPs array will be used to identify novel candidate set of predictive markers.
Genetic: Protein expression analysis — Tissue microarray made from formalin-fixed paraffin-embedded (FFPE) paired tumor and normal tissues is used for specific protein expression analysis by immunohistochemistry staining.

SUMMARY:
The goal of this laboratory research is to look for genetic and epigenetic markers that can predict which patients with stage III colorectal cancer will benefit from fluorouracil-based adjuvant chemotherapy.

DETAILED DESCRIPTION:
This is a prospective project in collecting and assessing clinical outcomes data related to molecular profiling of tumors based on samples from peripheral blood, primary tumor, and adjacent normal colorectal tissue.

Objectives:

1. Validation of predictive value of known markers CpG island methylator phenotype (CIMP) and microsatellite instability (MSI) in the response to 5-fluorouracil-based chemotherapy in patients with stage III colorectal cancer.
2. Exploratory evaluation of the potential predictive values of known genetic variations including, but not limited to, KRAS mutations, BRAF mutations, PIK3A mutations, and EGFR mutations, etc.
3. Exploratory identification and evaluation of the predictive value of novel methylation aberrations identified by whole-genome bisulfite sequencing.
4. Exploratory identification and evaluation of the predictive value of novel genetic aberrations discovered by RNA-sequencing (RNA-seq) or genome-wide association study (GWAS).

Outline:

Blood is collected at baseline and examined for single-nucleotide polymorphisms (SNPs) and expression level of specific gene. Tumor and corresponding normal tissue at surgical resection and assessed for gene methylations, mutations, and expressions.

ELIGIBILITY:
Inclusion Criteria:

1. Requirements for tumor parameters

   1. Histologically confirmed colorectal adenocarcinoma.
   2. Stage III disease (any pT, N1-2, M0).
   3. Tumors must have been curatively resected (R0).
   4. No evidence of residual involved lymph node disease or metastatic disease at the time of registration.
2. Requirements for patient characteristics

   1. Patient is ≥ 18 years of age on the day of consenting to the study.
   2. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1 at the time of screening.
   3. Fertile patients must use effective contraception.
   4. Patients must demonstrate ability to understand and the willingness to sign a written informed consent document.
   5. Patients must demonstrate ability to complete study questionnaires.
   6. Patients must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up.
3. Required initial laboratory values

   1. Leukocytes ≥ 3,000/mm^3
   2. Absolute neutrophil count ≥ 1,500/mm^3
   3. Platelet count ≥ 100,000/mm^3
   4. Creatinine ≤ 1.5 times upper limit of normal (ULN)
   5. Total Bilirubin ≤ 1.5 times ULN
   6. Aspartate aminotransferase (AST) ≤ 2.5 times ULN
   7. Alanine aminotransferase (ALT) ≤ 2.5 times ULN

Exclusion Criteria:

1. Patients with a known history of allergic reactions attributed to compounds of similar chemical or biologic composition to fluorouracil.
2. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection-requiring intravenous antibiotics, or psychological, familial, sociological, or geographical condition that would limit compliance with study requirements
3. Following cardiovascular conditions within the past 6 months: Myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia, cerebrovascular accident or transient ischemic attack, deep vein thrombosis, other significant thromboembolic event.
4. Known human immunodeficiency virus (HIV)-positive patients and those with known hepatitis B or C.
5. Patients with evidence of other primary malignancies within the past 5 years, excluding adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix.
6. Pregnant or nursing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed colorectal adenocarcinoma consecutively enrolled at the Department of Gastrointestinal Surgery II, Renmin Hospital, Wuhan University between Jan 2020 and Jan 2025.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to recurrence (TTR) | 3 years after surgery
  Time to any event, except non-cancer-related death. All recurrences, treatment-related deaths, second same or other primary cancers, and deaths from other cancers are considered to be events. Loss to follow-up and non-cancer-related deaths are censored. Associations between TTR and genetic and epigenetic markers will be analyzed.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 3 years, 5 years after surgery
  Time to any event, irrespective of cause. All events are included, except loss to follow-up. Associations between DFS and genetic and epigenetic markers will be analyzed.
Cancer-specific survival (CSS) | 3 years, 5 years after surgery
  Time to death caused by the same cancer, whether due to the original tumor or to a second primary same cancer. The only event is death from the same cancer, without taking into account whether the death is caused by the primary tumor or a second same cancer. Locoregional recurrence, distant metastases, second primary same cancers, and second other primary cancers are ignored. Deaths from other cancers, non-cancer-related deaths, treatment-related deaths, and loss to follow-up are censored. Associations between CSS and genetic and epigenetic markers will be analyzed.
Overall survival (OS) | 3 years, 5 years after surgery
  Time to death, irrespective of cause. There is no need to specify whether the death was due to cancer. Locoregional recurrence, distant metastases, second primary colorectal cancers, and second other primary cancers are ignored. Loss to follow-up is censored. Associations between OS and genetic and epigenetic markers will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastrointestinal Surgery II, Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jover R, Nguyen TP, Perez-Carbonell L, Zapater P, Paya A, Alenda C, Rojas E, Cubiella J, Balaguer F, Morillas JD, Clofent J, Bujanda L, Rene JM, Bessa X, Xicola RM, Nicolas-Perez D, Castells A, Andreu M, Llor X, Boland CR, Goel A. 5-Fluorouracil adjuvant chemotherapy does not increase survival in patients with CpG island methylator phenotype colorectal cancer. Gastroenterology. 2011 Apr;140(4):1174-81. doi: 10.1053/j.gastro.2010.12.035. Epub 2010 Dec 24. PMID 21185836
- [Background] Carethers JM, Smith EJ, Behling CA, Nguyen L, Tajima A, Doctolero RT, Cabrera BL, Goel A, Arnold CA, Miyai K, Boland CR. Use of 5-fluorouracil and survival in patients with microsatellite-unstable colorectal cancer. Gastroenterology. 2004 Feb;126(2):394-401. doi: 10.1053/j.gastro.2003.12.023. PMID 14762775
- [Background] Gamazon ER, Huang RS, Cox NJ, Dolan ME. Chemotherapeutic drug susceptibility associated SNPs are enriched in expression quantitative trait loci. Proc Natl Acad Sci U S A. 2010 May 18;107(20):9287-92. doi: 10.1073/pnas.1001827107. Epub 2010 May 4. PMID 20442332
- [Background] Dai J, Gu J, Huang M, Eng C, Kopetz ES, Ellis LM, Hawk E, Wu X. GWAS-identified colorectal cancer susceptibility loci associated with clinical outcomes. Carcinogenesis. 2012 Jul;33(7):1327-31. doi: 10.1093/carcin/bgs147. Epub 2012 Apr 12. PMID 22505654
- [Background] Xing J, Myers RE, He X, Qu F, Zhou F, Ma X, Hyslop T, Bao G, Wan S, Yang H, Chen Z. GWAS-identified colorectal cancer susceptibility locus associates with disease prognosis. Eur J Cancer. 2011 Jul;47(11):1699-707. doi: 10.1016/j.ejca.2011.02.004. Epub 2011 Mar 12. PMID 21402474
- [Background] Lin M, Gu J, Eng C, Ellis LM, Hildebrandt MA, Lin J, Huang M, Calin GA, Wang D, Dubois RN, Hawk ET, Wu X. Genetic polymorphisms in MicroRNA-related genes as predictors of clinical outcomes in colorectal adenocarcinoma patients. Clin Cancer Res. 2012 Jul 15;18(14):3982-91. doi: 10.1158/1078-0432.CCR-11-2951. Epub 2012 Jun 1. PMID 22661538
- [Background] O'Donnell PH, Stark AL, Gamazon ER, Wheeler HE, McIlwee BE, Gorsic L, Im HK, Huang RS, Cox NJ, Dolan ME. Identification of novel germline polymorphisms governing capecitabine sensitivity. Cancer. 2012 Aug 15;118(16):4063-73. doi: 10.1002/cncr.26737. Epub 2012 Jan 3. PMID 22864933
- [Background] Yoon HH, Tougeron D, Shi Q, Alberts SR, Mahoney MR, Nelson GD, Nair SG, Thibodeau SN, Goldberg RM, Sargent DJ, Sinicrope FA; Alliance for Clinical Trials in Oncology. KRAS codon 12 and 13 mutations in relation to disease-free survival in BRAF-wild-type stage III colon cancers from an adjuvant chemotherapy trial (N0147 alliance). Clin Cancer Res. 2014 Jun 1;20(11):3033-43. doi: 10.1158/1078-0432.CCR-13-3140. Epub 2014 Mar 31. PMID 24687927
- [Background] Roepman P, Schlicker A, Tabernero J, Majewski I, Tian S, Moreno V, Snel MH, Chresta CM, Rosenberg R, Nitsche U, Macarulla T, Capella G, Salazar R, Orphanides G, Wessels LF, Bernards R, Simon IM. Colorectal cancer intrinsic subtypes predict chemotherapy benefit, deficient mismatch repair and epithelial-to-mesenchymal transition. Int J Cancer. 2014 Feb 1;134(3):552-62. doi: 10.1002/ijc.28387. Epub 2013 Sep 13. PMID 23852808
- [Background] Dalerba P, Sahoo D, Paik S, Guo X, Yothers G, Song N, Wilcox-Fogel N, Forgo E, Rajendran PS, Miranda SP, Hisamori S, Hutchison J, Kalisky T, Qian D, Wolmark N, Fisher GA, van de Rijn M, Clarke MF. CDX2 as a Prognostic Biomarker in Stage II and Stage III Colon Cancer. N Engl J Med. 2016 Jan 21;374(3):211-22. doi: 10.1056/NEJMoa1506597. PMID 26789870
- [Background] Sinicrope FA, Mahoney MR, Smyrk TC, Thibodeau SN, Warren RS, Bertagnolli MM, Nelson GD, Goldberg RM, Sargent DJ, Alberts SR. Prognostic impact of deficient DNA mismatch repair in patients with stage III colon cancer from a randomized trial of FOLFOX-based adjuvant chemotherapy. J Clin Oncol. 2013 Oct 10;31(29):3664-72. doi: 10.1200/JCO.2013.48.9591. Epub 2013 Sep 9. PMID 24019539
- [Background] Sinicrope FA, Shi Q, Smyrk TC, Thibodeau SN, Dienstmann R, Guinney J, Bot BM, Tejpar S, Delorenzi M, Goldberg RM, Mahoney M, Sargent DJ, Alberts SR. Molecular markers identify subtypes of stage III colon cancer associated with patient outcomes. Gastroenterology. 2015 Jan;148(1):88-99. doi: 10.1053/j.gastro.2014.09.041. Epub 2014 Oct 8. PMID 25305506
- [Background] Toiyama Y, Hur K, Tanaka K, Inoue Y, Kusunoki M, Boland CR, Goel A. Serum miR-200c is a novel prognostic and metastasis-predictive biomarker in patients with colorectal cancer. Ann Surg. 2014 Apr;259(4):735-43. doi: 10.1097/SLA.0b013e3182a6909d. PMID 23982750
- [Background] Calon A, Lonardo E, Berenguer-Llergo A, Espinet E, Hernando-Momblona X, Iglesias M, Sevillano M, Palomo-Ponce S, Tauriello DV, Byrom D, Cortina C, Morral C, Barcelo C, Tosi S, Riera A, Attolini CS, Rossell D, Sancho E, Batlle E. Stromal gene expression defines poor-prognosis subtypes in colorectal cancer. Nat Genet. 2015 Apr;47(4):320-9. doi: 10.1038/ng.3225. Epub 2015 Feb 23. PMID 25706628
- [Background] Kap EJ, Seibold P, Scherer D, Habermann N, Balavarca Y, Jansen L, Zucknick M, Becker N, Hoffmeister M, Ulrich A, Benner A, Ulrich CM, Burwinkel B, Brenner H, Chang-Claude J. SNPs in transporter and metabolizing genes as predictive markers for oxaliplatin treatment in colorectal cancer patients. Int J Cancer. 2016 Jun 15;138(12):2993-3001. doi: 10.1002/ijc.30026. Epub 2016 Feb 19. PMID 26835885
- [Background] Dienstmann R, Vermeulen L, Guinney J, Kopetz S, Tejpar S, Tabernero J. Consensus molecular subtypes and the evolution of precision medicine in colorectal cancer. Nat Rev Cancer. 2017 Mar 23;17(4):268. doi: 10.1038/nrc.2017.24. No abstract available. PMID 28332502
- [Background] Punt CJ, Buyse M, Kohne CH, Hohenberger P, Labianca R, Schmoll HJ, Pahlman L, Sobrero A, Douillard JY. Endpoints in adjuvant treatment trials: a systematic review of the literature in colon cancer and proposed definitions for future trials. J Natl Cancer Inst. 2007 Jul 4;99(13):998-1003. doi: 10.1093/jnci/djm024. Epub 2007 Jun 27. PMID 17596575